CLINICAL TRIAL: NCT05607667
Title: Efficacy and Safety of the J-Valve Transcatheter Aortic Valve Replacement System in Patients With Aortic Stenosis Disease
Brief Title: Clinical Trial in China for Aortic Valve Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Genesis Medtech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S202112-01
Record Dates: First submitted 2022-10-27; First posted 2022-11-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Diseases of Aortic Valve; Aortic Stenosis Disease
MeSH Terms: conditions — Aortic Valve Disease | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Treatment (Experimental): Device: J-Valve® valve delivery system， Transvascularized biological aortic valve system
  Interventions: Device: Transcatheter aortic valve replacement

INTERVENTIONS:
Device: Transcatheter aortic valve replacement — Transcatheter aortic valve replacement system

SUMMARY:
The purpose of this clinical study is to evaluate the effectiveness and safety of the transcatheter aortic valve system in the treatment of patients with severe aortic stenosis disease who are at high or prohibitive surgical risk.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, single-arm, clinical study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65;
2. Patients with symptomatic aortic valve regurgitation diseases, and New York Heart Association (NYHA) ≥ II;
3. Subject must have Society of Thoracic Surgeons (STS) score ≥8% or have been evaluated as inoperable by the surgical team [defined as rate of death #50% within 30 d post-surgery or accompanied with irreversible occasions of other factors prevent surgeries (such as heavily calcified (porcelain) ascending aorta, weakness, chest malformation, liver dysfunction, pulmonary dysfunction and so on ); (Note: age of inoperable patients can be expanded to ≥ 50);
4. Aortic valve anatomy is suitable for TAVR evaluated by the investigators;
5. Patients who can sign informed consent form, and are willing to accept relevant examinations and clinical follow-ups.

Exclusion Criteria:

1. Active endocarditis;
2. Acute myocardial infarction or coronary revascularization occurred within 1 month before procedure;
3. Cerebrovascular accident (CVA) occurred within 30 days before procedure;
4. The echocardiogram indicates the presence of mass, thrombus or vegetation in left ventricle and left atrium;
5. Hypertrophic obstructive cardiomyopathy;
6. Other valve diseases that need interventions;
7. Previous aortic valve implantation (mechanical or biological);
8. Allergic to Nickel-titanium alloys or contrast agents or cattle-originated products;
9. Known allergy or contraindication to all anticoagulation, or anticoagulation can not be used during the TAVR;
10. In presence one of the following (from selection to the day of procedure index): a other diseases that may shorten life expectancy to less than 12 months (recurrent or metastatic cancer, congestive heart failure); b drug abuse (such as cocaine, heroin and so on); c planned additional operations that may result in incompliance or data confusion;
11. Stenosis of common carotid artery, internal carotid artery or vertebral artery #70%;
12. Severe left ventricular dysfunction, left ventricular ejection fraction (LVEF) <20%;
13. Hepatic encephalopathy or acute active hepatitis;
14. Receiving hemodialysis;
15. Bleeding tendency or history of coagulopathy or refuse to receive transfusion;
16. Active gastrointestinal (GI) ulcer or bleeding;
17. Severe dementia;
18. Patients who need emergency surgery for any reason;
19. Patients are participating in other drugs or medical devices clinical trial;
20. Pregnant or plan to be pregnant, or are taking estrogen or estrogen-like drugs (Women suspected of pregnancy must have a negative serum or urine test for human villous gonadotropin prior to enrollment in the study);
21. Other inappropriate occasions according to the investigators.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-03 (Actual)

PRIMARY OUTCOMES:
Cumulative all-cause mortality | 12 months
  All-cause mortality within 12 months of TAVR procedure

SECONDARY OUTCOMES:
Device success | 30 days
  No operative death;The instrument was placed in the correct anatomical position, and the delivery assembly was successfully entered and withdrawn;No device-related surgical or interventional intervention (other than permanent pacemaker implantation)
Procedural success | : immediate post-surgical
  Technical success,No death,No device-related surgical or interventional intervention (except permanent pacemaker implantation),The artificial aortic valve achieved the expected value (mean transaortic pressure difference < 20mmHg or transaortic flow velocity < 3m/s; No moderate or greater artificial aortic regurgitation or perivalvular leakage)
Evaluation of bioprosthetic valve and cardiac function Evaluation of bioprosthetic valve and cardiac function Evaluation of bioprosthetic valve and cardiac function | 30 days, 6 months, 12 months
  Echocardiography was used to evaluate aortic valve function and cardiac function
Functional Improvement of heart ( NYHA） | 30 days, 6 months, 12 months
  NYHA classification of cardiac function was evaluated after operation
Quality of life（KCCQ） | 30 days, 6 months, 12 months
  Evaluation of postoperative Quality of life score improvement (KCCQ)
Major cardiovascular and cerebrovascular adverse events (MACCE) | before discharge/7days, 30 days, 6 months, 12 months
  Major adverse cardiovascular and cerebrovascular events (MACCE) included mortality, stroke, myocardial infarction, reoperation, arrhythmia, and conduction block.
Myocardial infarction | before discharge/7days, 30 days, 6 months, 12 months
  Incidence of myocardial infarction
Stroke | before discharge/7days, 30 days, 6 months, 12 months
  Grades include ischemic stroke (including transient ischemic attack, TIA) and hemorrhagic stroke Grades included ischemic stroke (including transient ischemic attack, TIA) and hemorrhagic stroke; Definitions included disabling stroke (modified Rankin score ≥2 at 90 days after stroke with an increase of >1 point) and nondisabling stroke (modified Rankin score <2 at 90 days after stroke with no increase in score). Stroke events should be recorded and the causes analyzed in detail.
Major bleeding (life-threatening or crippling) | before discharge/7days, 30 days, 6 months, 12 months
  Severe bleeding: BARC bleeding was defined as type 3a and above
Acute kidney injury | before discharge/7days, 30 days, 6 months, 12 months
  The incidence of AKIN stage 2 and above events was recorded.
Conduction block and malignant arrhythmia | before discharge/7days, 30 days, 6 months, 12 months
  The incidence of conduction block and malignant arrhythmias
Permanent pacemaker implantation | before discharge/7days, 30 days, 6 months, 12 months
  Permanent pacemaker implantation rate
TAVI related complications | before discharge/7days, 30 days, 6 months, 12 months
  These include conversion to surgery, accidental mechanical cardiopulmonary assistance, coronary occlusion, ventricular septal perforation, mitral valve damage or loss of function, cardiac tamponade, endocarditis, valve thrombosis, valve ectopic (displacement, embolization, misrelease), aortic dissection, aortic root rupture, and peripheral vascular complications.
Device defects | intraoperative
  Incidence of device defects
The incidence of adverse events The incidence of adverse events | 12 months
  Incidence of adverse events
The incidence of serious adverse events | 12 months
  Incidence of serious adverse events

CONTACTS AND LOCATIONS:
Locations (15):
- China (15):
  - Beijing Anzhen Hospital,Capital Medical University, Beijing
  - Chinese PLA General Hoapital, Beijing
  - Peking University Third Hospital, Beijing
  - Xuanwu Hospital Capital Medical University, Beijing
  - Xinqiao Hospital Army Medical Univer Sity, Chongqing
  - Guangdong Academy of Medical Sciences, Guangdong
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongshan Hospital, Shanghai
  - WEST CHINA hospital, Sichuan
  - The First Affiliated of Soochow University, Suzhou
  - Xijing Hospital of the Fourth Military Medical University, Xi'an
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen
  - Fuwai Yunnan Cardiovascular Hospital, Yunnan
  - The Second Affiliated Hospital of Zhejiang University, Zhangjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No